CLINICAL TRIAL: NCT03067987
Title: Safety and Efficacy of Low Intensity Shockwave for the Treatment of Erectile Dysfunction- Comparison of Two Treatment Schedule
Brief Title: Safety and Efficacy of Low Intensity Shockwave for the Treatment of Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: DIREX SYSTEMS CORPORATION (Industry)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Urologist/ Director of Male Reproductive Medicine/ Assistant professor Urology Department University of Miami, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160335
Record Dates: First submitted 2017-02-23; First posted 2017-03-01 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Vasculogenic Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 720 shockwave therapy (Active Comparator): 5 daily sessions of shockwave therapy within a week (Monday, Tuesday, Wednesday, Thursday, Friday), in which 720 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura).
  Interventions: Device: Low Intensity Linear Shockwave Device for the Treatment of Erectile Dysfunction.
- 600 shockwave therapy (Active Comparator): Three sessions of shockwave therapy per week (Monday, Wednesday, Friday) for 2 consecutive weeks, in which 600 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura)
  Following the last treatment session, each patient will resume his baseline consumption of phosphodiesterase 5 inhibitor, in terms of type and dose of drug, for the remainder of study duration.
  Interventions: Device: Low Intensity Linear Shockwave Device for the Treatment of Erectile Dysfunction.

INTERVENTIONS:
Device: Low Intensity Linear Shockwave Device for the Treatment of Erectile Dysfunction. — This is a prospective, randomized, clinical study aimed to evaluate the safety and efficacy of the two treatment schedules on symptomatic erectile dysfunction patients. The patients are randomized in a 1:1 ratio into two active treatment groups.
  Group A: 5 daily sessions within a week (Monday, Tuesday, Wednesday, Thursday, Friday), in which 720 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura).
  Group B: Three sessions per week (Monday, Wednesday, Friday) for 2 consecutive weeks, in which 600 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura)
  .
  Other Names: RENOVA-ED

SUMMARY:
Renova- Erectile Dysfunction (ED) is a Linear Shockwaves (LISW) device which incorporates a unique shockwave transducer operable to deliver shockwaves to a treated region. Shockwaves are aimed at the left and right corpora cavernosa and the crura. The study is aimed at determining the safety and effectiveness of this new type LISW in the relief of erectile dysfunction.

HYPOTHESIS Alternate Hypothesis (HA): Active Treatment groups will show a >2-point increase in the IIEF-EF score from baseline for mild erectile dysfunction, and >5 points for moderate erectile dysfunction and will show significant change.

Null Hypothesis (HO): There is no difference from baseline and after-treatment in Treatment groups for alleviating erectile dysfunction measured using International Index of Erectile Function score (IIEF-EF).

Primary Efficacy Objective: To evaluate change of International Index of Erectile Function score Questionnaire score from baseline to follow-ups 1, 3 and 6 months' post treatment.

Secondary Objectives:To study sexual activity improvement leading to optimal penetration at follow-ups according to:

* SEP- Sexual Encounter Profile Questionnaire.
* GAQ- Global Assessment Questionnaire.
* EHS- Erection Hardness Score.

DETAILED DESCRIPTION:
Renova-Erectile dysfunction (ED) is a Linear Shockwaves (LISW) device which incorporates a unique shockwave transducer operable to deliver shockwaves to a treated region confined to a narrow rectangle. Shockwaves generation follows the electromagnetic principle.

Linear Shockwaves (LISW), as a treatment for erectile dysfunction has been in evaluation in contemporary medicine, It has been in use for the last three years.

The present study is about a device called "Renova-erectile dysfunction", in which shockwaves are focused onto line segments for improved organ coverage. Shockwaves produced by "Renova-erectile dysfunction" are aimed at the left and right corpora cavernosa and the crura. The study is aimed at determining the safety and effectiveness of this new type LISW in the relief of erectile dysfunction.

Rationale:Linear Shockwaves has been known to bolster angiogenesis by increasing the levels of vascular endothelial growth factor.

Principal mode of action used in other disease:

* Coronary Artery Disease: Kikuchi et al.3 showed significantly improved symptoms and decreased nitroglycerin use in patient who had a coronary artery bypass grafting and were suffering from stable angina.
* Bone Healing: Haupt et al.4 showed that Low intensity shock waves treated group showed radiological signs of faster healing.
* Calcifying tendinitis: Rompe et al.5 showed that shock wave to patient suffering from calcifying tendinitis showed a 62.5% partial and complete disintegration of the the deposits. Moreover, 85% of the patients reported improvement at 24-week follow up period.
* Diabetic Foot Ulcers: Wang et al.6 showed that Extracorporeal Shock Wave Therapy (ESWT) to patients with diabetic foot ulcer showed complete improvement in 31% and partial improvement in 58%.Moreover,Extracorporeal Shock Wave Therapy showed significantly better clinical results and local blood flow perfusion, higher cell concentration, and activity than the Hyperbaric Oxygen group.

Preliminary Studies:

Contemporary literature shows two important studies in this field both conducted by Verdi et al.

The efficacy trial study published in 2010 recruited 20 men with vasculogenic erectile dysfunction and were given serial 2 sessions of treatment for about 3 weeks followed by 3 - week no intervention period. At 1-month duration there was a significant improvement in their erectile function measured by International Index of Erectile Function domain scores (20.9 5.8 vs 13.5 4.1, p < 0.001). This significant result was consistent at 6-month follow up. Moreover, no pain or adverse event was noted during the follow-up period.

The second randomized, double-blind, sham controlled study by showed that treatment group showed better outcome than control group measured using International Index of Erectile Function-Erectile Function domain (mean square root of sample size 6.7 0.9 vs 3.0 1.4, p 0.0322) at the first follow-up. Additionally, penile hemodynamics improve significantly in the treatment group in comparison to control group (maximal post-ischemic penile blood flow 8.2 vs 0.1 ml per minute per dl, p 0.0001).

Primary Efficacy Objective:To evaluate change of Erectile Function-Erectile Function score 9 from baseline to follow-ups 1, 3 and 6 months' post treatment.

Secondary Objectives:To study sexual activity improvement leading to optimal penetration at follow-ups according to:

* SEP- Sexual Encounter Profile.
* GAQ- Global Assessment Questions.
* EHS- Erection Hardness Score.

STUDY DESIGN Accrual goal: A total of 80 patients with Vasculogenic erectile dysfunction meeting the eligibility criteria will be recruited from the Department of Urology clinic.

Duration of Study Participation: The total duration of the study will be for 7 months- including 1-month pretreatment (washout) followed by a period of 6 months' follow-up after the treatment.

Screening Evaluations and Procedures: The first visit of the patients will be for screening and medical evaluation. Patient's medical co-medication history will be collected and documented and a physical examination will be performed.

Previous month's blood test results will be reviewed including a general chemistry panel, a lipid profile, hemoglobin A1C and testosterone levels during chart review.

Patients will sign an informed consent and will answer the Erectile Function-Erectile Function questionnaire to see if they fit the criteria for enrollment. In case they meet all inclusion criteria (and do not meet any exclusion criteria), they will be recruited to the study.

Patients who have been using phosphodiesterase 5 inhibitor (PDE5-i) in the last 4 weeks will report on their medicine type and dosage, and this data will be recorded in their files (reported prior to consent and gathered from chart review).

Pre-Treatment Procedures and Evaluations : Upon evaluating the inclusion/exclusion criteria, patients will be recruited to the study and randomized into one of the two groups in a 1:1 ratio (randomization will be performed by a computer software maintained by the Department of Urology). Patients randomized to the treatment groups will be instructed to stop any use of phosphodiesterase 5 inhibitor for 4 weeks prior to first treatment session and refrain from using any other erectile dysfunction therapy option during the study. They will be instructed to undergo a phosphodiesterase 5 inhibitor washout period of 4 weeks prior to treatment and to avoid using phosphodiesterase 5 inhibitor or any other erectile dysfunction treatment during the entire study duration (shockwave treatment and follow-ups). After the washout period and before the first treatment session, patients will answer the IIEF-EF, SEP and EHS questionnaires for baseline evaluation.

Treatment procedure: The treatment session lasts approximately 20 minutes and may be performed in an office environment. Treatment is applied in the physician's office. For session and treatment details (see below)

During the treatment, the same total number of shocks will be delivered according to the two treatment schedules as follows:

Group A:

5 daily sessions within a week (Monday, Tuesday, Wednesday, Thursday, Friday (MTWThF), in which 720 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura).

Group B:

Three sessions per week Monday, Wednesday, Friday (MWF) for 2 consecutive weeks, in which 600 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura)

Following the last treatment session, each patient will resume his baseline consumption of phosphodiesterase 5 inhibitor, in terms of type and dose of drug, for the remainder of study duration.

Follow-Up Procedures and Evaluations:Follow-up visits will be conducted at month 1, month 3 and month 6 after the last treatment session and shall include:

Measuring IIEF-EF, GAQ, SEP, and EHS scores of patients at the clinic at every follow-up visit

Reporting and recording adverse events at every follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be willing and able to provide informed consent.
* The patient is a male between >30 and <80 years of age.
* PDE5i responsive or non-responsive. If on PDE5i patient will discontinue medication for 4 weeks before IIEF.
* Stable sexual relationship for over 3 months prior to enrollment.
* A minimum of 2 sexual attempts per month for at least one month prior to enrollment.
* Erectile dysfunction lasting for over 6 months and not more than 5 years.
* Baseline IIEF-EF score between 11 and 25. If taking PDE5i, stop medication for at least 4 weeks before baseline IIEF-EF.
* Testosterone level 300-1000 ng/dL.
* If diabetic, HgbA1C level ≤ 7.5% within 1 month prior to enrollment.

Exclusion Criteria:

* The patient is currently or has participated in another study within the past three months, that may interfere with the results or conclusions of this study.
* The patient is under judicial protection (prison or custody).
* The patient is an adult under guardianship.
* The patient refuses to sign the consent.
* History of radical prostatectomy or extensive pelvic surgery ever.
* Past radiation therapy of the pelvic region within 12 months prior to enrollment.
* Recovering from any cancer within 12 months prior to enrollment.
* Neurological disease such as Alzheimers or Parkinsons disease which affects erectile function at the discretion of the investigator.
* Psychiatric diagnosis or medications such as antidepressants which affects erectile function or any other medications at the discretion of the investigator.
* Anatomical malformation of the penis, including Peyronie's disease.
* Testosterone level <300 or >1000 ng/dL within 1 month prior to enrollment.
* HgbA1C level > 7.5% within 1 month prior to enrollment.
* Androgen deprivation treatment in the last year.
* History of spinal cord injury.
* The patient is taking blood thinners (eg Coumadin, Plavix)

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulhall JP. Defining and reporting erectile function outcomes after radical prostatectomy: challenges and misconceptions. J Urol. 2009 Feb;181(2):462-71. doi: 10.1016/j.juro.2008.10.047. Epub 2008 Dec 13. PMID 19084865
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Vardi Y, Appel B, Kilchevsky A, Gruenwald I. Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study. J Urol. 2012 May;187(5):1769-75. doi: 10.1016/j.juro.2011.12.117. Epub 2012 Mar 15. PMID 22425129
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Wang CJ, Kuo YR, Wu RW, Liu RT, Hsu CS, Wang FS, Yang KD. Extracorporeal shockwave treatment for chronic diabetic foot ulcers. J Surg Res. 2009 Mar;152(1):96-103. doi: 10.1016/j.jss.2008.01.026. Epub 2008 Mar 7. PMID 18619622
- [Background] Rompe JD, Rumler F, Hopf C, Nafe B, Heine J. Extracorporal shock wave therapy for calcifying tendinitis of the shoulder. Clin Orthop Relat Res. 1995 Dec;(321):196-201. PMID 7497669
- [Background] Haupt G, Haupt A, Ekkernkamp A, Gerety B, Chvapil M. Influence of shock waves on fracture healing. Urology. 1992 Jun;39(6):529-32. doi: 10.1016/0090-4295(92)90009-l. PMID 1615601
- [Background] Kikuchi Y, Ito K, Ito Y, Shiroto T, Tsuburaya R, Aizawa K, Hao K, Fukumoto Y, Takahashi J, Takeda M, Nakayama M, Yasuda S, Kuriyama S, Tsuji I, Shimokawa H. Double-blind and placebo-controlled study of the effectiveness and safety of extracorporeal cardiac shock wave therapy for severe angina pectoris. Circ J. 2010 Mar;74(3):589-91. doi: 10.1253/circj.cj-09-1028. Epub 2010 Feb 4. PMID 20134096
- [Background] Melman A, Gingell JC. The epidemiology and pathophysiology of erectile dysfunction. J Urol. 1999 Jan;161(1):5-11. PMID 10037356
- [Background] Vlachopoulos C, Rokkas K, Ioakeimidis N, Aggeli C, Michaelides A, Roussakis G, Fassoulakis C, Askitis A, Stefanadis C. Prevalence of asymptomatic coronary artery disease in men with vasculogenic erectile dysfunction: a prospective angiographic study. Eur Urol. 2005 Dec;48(6):996-1002; discussion 1002-3. doi: 10.1016/j.eururo.2005.08.002. Epub 2005 Aug 24. PMID 16174548
- [Derived] Katz JE, Molina ML, Clavijo R, Prakash NS, Ramasamy R. A Phase 2 Randomized Trial To Evaluate Different Dose Regimens of Low-intensity Extracorporeal Shockwave Therapy for Erectile Dysfunction: Clinical Trial Update. Eur Urol Focus. 2018 Apr;4(3):336-337. doi: 10.1016/j.euf.2018.07.011. Epub 2018 Jul 17. PMID 30025713

RESULTS

PARTICIPANT FLOW:
Groups:
- 600 Shockwave Therapy: Three sessions of shockwave therapy per week (Monday, Wednesday, Friday) for 2 consecutive weeks, in which 600 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura)
Period: Overall Study
Arm/Group | 720 Shockwave Therapy | 600 Shockwave Therapy
Started | 50 | 53
Completed | 40 | 40
Not Completed | 10 | 13
Not completed — Lost to Follow-up | 7 | 10
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 720 Shockwave Therapy | 600 Shockwave Therapy | Total
Number analyzed (Participants) | 50 | 53 | 103
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [30 to 80] | 52 [30 to 80] | 52.25 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 50 | 53 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 23 | 47
  Not Hispanic or Latino | 26 | 30 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 5 | 2 | 7
  Black or African American | 17 | 20 | 37
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: International Index of Erectile Function (IIEF-EF) Questionnaire
Description: IIEF is a 15 item self-administered questionnaire assessing erectile dysfunction and treatment outcomes. Total IIEF score range from 5-25 with scores classifying erectile dysfunction (ED) as: severe (5-7); moderate (8-11); mild to moderate (12-16); mild (17-21) and no ED (22-25). The questionnaire will be assessed at baseline (before 1 month washout prior to treatment initiation), 1 month follow up (at 2 months), 3 month follow up (at 4 months) and 6 months follow up (at 7 months).
  Time Frame: 7 months
Time Frame: 7 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 720 Shockwave Therapy | 600 Shockwave Therapy
Number analyzed (Participants) | 40 | 40
score on a scale
  SCORE AT BASELINE | 18 [11 to 25] | 17.9 [11 to 25]
  SCORE AT 1 MONTHS | 20.5 [11 to 25] | 19.7 [11 to 25]
  SCORE AT 3MONTHS | 19.8 [11 to 25] | 21.2 [11 to 25]
  SCORE AT 6 MONTHS | 20.9 [11 to 25] | 21.4 [11 to 25]
Statistical Analysis 1: Comparison: 720 Shockwave Therapy vs 600 Shockwave Therapy; Test type: Superiority; p < 0.007, ANOVA

2. Secondary Outcome: Erection Hardness Score (EHS)
Description: EHS rates the hardness of erection on a scale of 1-4 assessed at baseline (before 1 month washout prior to treatment initiation), 1 month follow up (at 2 months), 3 month follow up (at 4 months) and 6 months follow up (at 7 months). A score of 0 = penis does not enlarge; 1 = penis is larger but not hard; 2 = penis is hard but not hard enough for penetration; 3 = penis is hard enough for penetration but not completely hard; 4 = penis is completely hard and fully rigid.
Time Frame: 7 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | 720 Shockwave Therapy | 600 Shockwave Therapy
Number analyzed (Participants) | 40 | 40
score on a scale
  SCORE AT BASELINE | 2.5 [0 to 4] | 2.7 [0 to 4]
  SCORE AT 1 MONTH | 3.1 [0 to 4] | 3 [0 to 4]
  SCORE AT 3 MONTHS | 3.1 [0 to 4] | 3 [0 to 4]
  SCORE AT 6 MONTHS | 3.1 [0 to 4] | 3.2 [0 to 4]
Statistical Analysis 1: Comparison: 720 Shockwave Therapy vs 600 Shockwave Therapy; Test type: Superiority; p = 0.0006, ANOVA

3. Secondary Outcome: Sexual Encounter Profile (SEP)
Description: Sexual Encounter Profile (SEP) is a measure of efficacy of erectile dysfunction therapy. Improved responses to treatment will be reported as the percentage of participants that responds "yes" and non-improvement responses to treatment will be reported as the percentage of participants that responds "no".
Time Frame: 7 months
Measure: Number; unit: percentage of participants
Arm/Group | 720 Shockwave Therapy | 600 Shockwave Therapy
Number analyzed (Participants) | 40 | 40
percentage of participants
  SEP-Q2 (YES) | 96 | 95
  SEP-Q2 (NO) | 4 | 5
  SEP-Q3 (YES) | 69 | 70
  SEP-Q3 (NO) | 31 | 30

4. Secondary Outcome: Global Assessment Question (GAQ)
Description: Global Assessment Question (GAQ) is a measure of perceived improvements in erectile function and sexual ability. Improved responses to treatment will be reported as the percentage of participants that responds "yes" and non-improvement responses to treatment will be reported as the percentage of participants that responds "no".
Time Frame: 7 months
Measure: Number; unit: percentage of participants
Arm/Group | 720 Shockwave Therapy | 600 Shockwave Therapy
Number analyzed (Participants) | 40 | 40
percentage of participants
  GAQ-Q1 (YES) | 52 | 53
  GAQ-Q1 (NO) | 48 | 47
  GAQ-Q2 (YES) | 74 | 73
  GAQ-Q2(NO) | 26 | 27

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 720 Shockwave Therapy | 600 Shockwave Therapy
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/53
Other Adverse Events (participants affected / at risk) | 0/50 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03067987/Prot_SAP_000.pdf